CLINICAL TRIAL: NCT04181346
Title: Phase II Study of Pregabalin for the Prevention of Chemotherapy Induced Nausea and Vomiting
Brief Title: Pregabalin for the Prevention of Chemotherapy Induced Nausea and Vomiting
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Felipe Melo Cruz, PhD, Head of Medical Oncology Department, Faculdade de Medicina do ABC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBCC 01
Record Dates: First submitted 2019-11-22; First posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Nausea
Keywords: pregabalin; nausea
MeSH Terms: conditions — Nausea | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: chemotherapy-naive patients, scheduled to receive moderately and highly emetogenic chemotherapy will be randomized for two arms: pregabalin and placebo.
  All patients received will receive IV ondansetron 8 mg, dexamethasone 10 mg and ranitidine 50 mg before chemotherapy on day 1 and oral dexamethasone 4 mg, bd, on days 2 and 3.
Who Masked: Participant, Investigator
Masking Description: double blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin (Experimental): Pregabalin 75mg, twice a day, from the night before chemotherapy to day 5
  Interventions: Drug: Pregabalin
- Placebo (Experimental): Placebo, twice a day, from the night before chemotherapy to day 5
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — antipsychotic
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
phase II randomized, double-blind, placebo-controlled trial to investigate whether pregabalin can improve the complete control of nausea and vomiting (primary end point)

DETAILED DESCRIPTION:
chemotherapy-naive patients, scheduled to receive moderately and highly emetogenic chemotherapy.

All patients will receive IV ondansetron 8 mg, dexamethasone 10 mg and ranitidine 50 mg before chemotherapy on day 1 and oral dexamethasone 4 mg, bd, on days 2 and 3.

Patients will be randomly assigned to take pregabalin 75 mg or placebo, bd, from the night before chemotherapy to day 5.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to receive their first cycle of moderately to highly emetogenic chemotherapy;
* 18 years or older;
* Eastern Cooperative Oncology Group < 2

Exclusion Criteria:

* Nausea or vomiting 24h before randomization
* aspartate aminotransferase / alanine aminotransferase above 3 times the upper limit
* Severe cognitive compromise;
* regular use of corticosteroids, opioid, benzodiazepines, tricyclic antidepressant, or cannabinoids within 30 days before randomization;
* brain metastasis;
* chronic alcoholism;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving complete control of nausea and vomiting | five days

CONTACTS AND LOCATIONS:
Locations (1):
- IBCC Oncologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No